CLINICAL TRIAL: NCT07192679
Title: MAGNIFY - Pulmonary Magnetic Resonance Imaging for Cystic Fibrosis
Acronym: MAGNIFY
Status: Recruiting | Type: Observational
Sponsor: Sheffield Teaching Hospitals NHS Foundation Trust (Other)
Collaborators: University of Sheffield (Other)
Responsible Party: Sponsor
Other Study IDs: STH22784
Record Dates: First submitted 2025-09-04; First posted 2025-09-25 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Cystic Fibrosis (CF)
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Cohort 1 - MMAVIC protocol: Twenty patients who previously participated in the MMAVIC study, eligible to be on the new regime of CF therapies. These patients will be recruited and invited to attend 4 visits over 3 years.
- Cohort 2: Patients not eligible for HEMT: A combination of approximately ten children and ten adults who are either not eligible to take HEMT or have not tolerated highly effective modulator treatment (HEMT). Previous MMAVIC participants not on HEMT are also eligible for this cohort. These patients will be invited to attend 3 visits over 2 years.
- Cohort 3: School-age children on standard of care treatment: Twenty children who are receiving the current standard of care treatment, including HEMT or other CFTR modulators. These patients will be invited to attend 2 visits - 1 year apart.
- Cohort 4: Pre-school children on standard of care treatment: Up to 20 children under the age of 5 years, who are receiving the current standard of care, including CFTR modulator therapies. These participants will have a single visit.

SUMMARY:
This research study is looking at new ways of measuring the function of the lungs in patients with cystic fibrosis. This study is using the most advanced methods for measuring lung function including 2 tests called hyperpolarised gas magnetic resonance imaging (HP MRI) and multiple breath washout (MBW), to better understand changes in the lungs over time.

HP MRI involves taking pictures of the air in your lungs after breathing in a harmless gas (xenon). MBW is a breathing test used to calculate something called the lung clearance index (LCI).

By measuring these tests on the same day, alongside standard lung function tests, we aim to understand lung function in greater detail than ever before.

ELIGIBILITY:
General Inclusion criteria

For eligibility into MAGNIFY, subjects should meet all of the following criteria:

1. A confirmed clinical diagnosis of CF, consisting of 2 confirmed disease-causing CFTR mutations along with either positive sweat chloride (>60mmol/L, measured before starting CFTR modulator therapy) or a clinical picture consistent with CF as judged by a senior CF physician. Patients will be under one of named regional CF centres above.
2. Be able to attend the local facility for scans (Royal Hallamshire Hospital, Sheffield).

For eligibility into 129Xe-MRI and lung function (cohort 1,2 and 3)

1. Aged 5 years and above
2. FEV1 >30% predicted (best in the previous 6 months) For eligibility for cohort 1

1. Previous participation in the MMAVIC study, with at least one prior visit where lung ventilation MRI was successfully measured.

For eligibility into cohort 4 for 1H MRI only:

1. Aged between 1 and 5 years of age

General Exclusion criteria

Patients who meet any of the following criteria will be excluded from the study. Further exclusions may be applied at the discretion of the principal investigators.

1. Previous lung transplant.
2. Infection with organisms of the Burkholderia cepacia complex, MRSA or Mycobacterium abscessus.
3. Pregnancy.
4. Resting SpO2 < 90% in room air.
5. Inability to comfortably lie supine for more than 60 minutes.
6. Any contraindication(s) to MRI scanning as per the MRI questionnaire used in clinical practice by the University of Sheffield MRI unit, Royal Hallamshire Hospital.

Research visit (temporary) exclusion criteria

1. Pulmonary exacerbation within 4 weeks as defined by no new treatments in that time, no clinically significant change in their symptoms or spirometry (as judged by attending physician).
2. Pregnancy. Patients who become pregnant prior to consent or during the study can remain in the study. However, no research visits will take place during pregnancy.

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Adults and children with cystic fibrosis
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2024-02-21 (Actual); Primary Completion 2028-01-01 (Estimated); Study Completion 2028-01-01 (Estimated)

PRIMARY OUTCOMES:
Ventilation defect percent (VDP) as measured by 129Xe-MRI | Up to 3 years, depending on cohort.
  The primary endpoint will be changes in the 129Xe-MRI metric; ventilation defect percent (VDP) between study visits.

SECONDARY OUTCOMES:
XeMRI outcome measures - Ventilation Heterogeneity Index | up to 3 years
  Similar analysis to the primary outcome will be conducted for Ventilation Heterogeneity Index (VHI)
XeMRI outcome measures - individual defects | up to 3 years
  Similar analysis to the primary outcome will be conducted for the number and size (single measure) of individual defects
XeMRI outcome measures - reversibility index | up to 3 years
  Similar analysis to the primary outcome will be conducted for reversibility index.
Lung function metrics - LCI | Up to 3 years
  Similar analysis will be conducted for the major lung function test metric - LCI, Scond, Sacin (from MBW).
  R5, R5-R20, X5 and Ax from AOS. RV/TLC from body plethysmography. FEV1, FEV1/FVC from spirometry.
Lung function metrics - Scond (from MBW). | Up to 3 years
  Similar analysis will be conducted for the major lung function test metric - Scond, an outcome marker measured from MBW that represents ventilation heterogeneity in the conducting airways within the lung.
  R5, R5-R20, X5 and Ax from AOS. RV/TLC from body plethysmography. FEV1, FEV1/FVC from spirometry.
Lung function metrics - Sacin (from MBW). | Up to 3 years
  Similar analysis will be conducted for the major lung function test metric - Sacin, an outcome marker measured from MBW that represents ventilation heterogeneity in the acinar airways within the lung.
  R5, R5-R20, X5 and Ax from AOS. RV/TLC from body plethysmography. FEV1, FEV1/FVC from spirometry.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Sheffield MRI Unit, Sheffield, United Kingdom

IPD SHARING:
Plan to Share IPD: No